CLINICAL TRIAL: NCT02714387
Title: Prospective Cohort of Patients Hospitalized in West French Intensive Care Units.
Brief Title: Non Traumatic Neuro-Vascular Diseases Critical Complications : a Prospective Cohort Study
Acronym: ATLANREA
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0207 cohorte fiche 1
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Non Traumatic Acute Brain Injury
Keywords: Non traumatic acute brain injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, peripheral blood mononuclear cells, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: Patients with Non Traumatic Neuro-Vascular Diseases. Medical data concerning ICU stay will be collected.
  Interventions: Other: Collection of medical data

INTERVENTIONS:
Other: Collection of medical data — A code will be applied to each patient included. Medical data such as demography, Simplified Acute Physiological Score II (SAPS II), Sequential Organ Failure Assessment (SOFA), procedures and complications during ICU stay will be collected.

SUMMARY:
The purpose of this observational epidemiological study is to investigate the management and the complications associated with Non Traumatic Neuro-Vascular Diseases. Data will be analysed to answer pre-defined scientific projects and to improve management of these conditions.

DETAILED DESCRIPTION:
Anonymous data will be collected by study coordinators in a secured e-database. Cross audit will be performed to check data.

ELIGIBILITY:
Inclusion Criteria:

* Non Traumatic Neuro-Vascular Diseases

Exclusion Criteria:

* Consent withdrawal

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in ICU for Non Traumatic Neuro-Vascular Diseases
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-02; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
in ICU stay complications | Within the first 28 days after ICU admission date
  Hospital acquired infections (epidemiology, risk factors, antibiotic susceptibility of pathogens), Organ failures (incidence, risks factors), Bleeding, Hemorrhage Intra-Cranial Hypertension, Brain Ischemia, Mechanical ventilation weaning, Extubation failure

SECONDARY OUTCOMES:
Duration in mechanical ventilation | in ICU (up to 90 days)
ICU length of stay | in ICU (up to 90 days)

OTHER OUTCOMES:
Death | in ICU (up to 180 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, PhD, MD, Study Chair
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - CHU de Brest La Cavale Blanche, Brest
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours